CLINICAL TRIAL: NCT02544789
Title: Phase II, Multi-center, and Pharmacokinetic Study of Efficacy, Safety and Pharmacokinetic of Clofarabine in Chinese Pediatric Patients With Refractory or Relapsed Acute Lymphoblastic Leukemia
Brief Title: Clofarabine in Chinese Pediatric Patients With Refractory or Relapsed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-3-C01
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- clofarabine (Experimental): Clofarabine (Betta Pharmaceuticals Co., Ltd, Zhejiang, China) was administered intravenously at 52 mg/m2 over 2 hours daily for 5 consecutive days. During the first two induction cycles, patients who did not achieve an objective response were taken off the study, and responsive patients continued to receive consolidation for a maximum 11 cycles if non-hematological toxicity was grade 2 or less.
  Interventions: Drug: Clofarabine

INTERVENTIONS:
Drug: Clofarabine — Clofarabine (Betta Pharmaceuticals Co., Ltd, Zhejiang, China) was administered intravenously at 52 mg/m2 over 2 hours daily for 5 consecutive days. During the first two induction cycles, patients who did not achieve an objective response were taken off the study, and responsive patients continued to receive consolidation for a maximum 11 cycles if non-hematological toxicity was grade 2 or less.

SUMMARY:
Outcomes for children with relapsed/refractory (R/R) acute lymphoblastic leukemia (ALL) are dismal. Therefore, the investigators performed this multicenter, phase II study to evaluate the efficacy and , safety and pharmacokinetic of clofarabine in Chinese pediatric patients with R/R ALL

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (younger than 21 years old) with acute lymphoblastic leukemia confirmed by histology
* Refractory or relapsed acute lymphocytic leukemia who had received at least two drugs treatment
* No prior chemotherapy within 2 weeks before entry and resolution of toxic effects from prior therapy
* Normal cardiac function, adequate hepatic function [total bilirubin ≤1.5× upper limit of normal (ULN), aspartate aminotransferase (AST) alanine aminotransferase (ALT) ≤ 3ULN] and renal function (serum creatinine ≤ 2 ULN)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy more than 3 months

Exclusion Criteria:

* AEs not recovered from prior therapy
* Within 3 months from allogeneic or autologous stem cell transplantation
* With central nervous involvement or uncontrolled infection
* Patients who used clofarabine before or allergic to fludarabine or cladribine

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-06; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
overall response rate | 8 weeks

SECONDARY OUTCOMES:
patients suffering adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jin Lu, MD, Study Chair — Department of Pediatrics, Peking University People's Hospital
Locations (6):
- China (6):
  - Department of Pediatrics, Peking University People's Hospital, Beijing
  - Department of Phase 1 Clinical Trial, Peking University People's Hospital, Beijing
  - Guangdong General Hospital, Guangdong Academy of Medical Science, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - The First Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou